CLINICAL TRIAL: NCT03325140
Title: Platelet Transfusion Efficacy in Critically Ill Patients
Brief Title: Platelet Transfusions in Critically Ill Patient
Acronym: RE-CCIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RE-CCIP (29BRC17.0157)
Record Dates: First submitted 2017-10-21; First posted 2017-10-30 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Platelet Transfusion; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Between 10 and 15% of critically ill patients require platelet transfusion within their intensive care unit (ICU).

Platelets (PLT) are given to prevent bleeding in thrombocytopenic patients or to treat bleeding as part of massive transfusion or in bleeding thrombocytopenic patients.

International and local guidelines (American Association of Blood Banks-AABB) are mainly based on experts' opinion. The efficacy of PLT transfusion in the ICU setting remains poorly studied and unknown and the administration of PLT may be associated with adverse effects including an increased risk of hospital acquired infection. Finally, the short PLT shelve-life may be responsible for inventory issues. Altogether, this makes very important to improve the evidence that support PLT transfusion in ICU patients.

This is a multicentre prospective observational study that aims to first determine PLT transfusion efficacy and to identify the parameters associated with transfusion efficacy and to analyse the compliance with international (and local) guidelines of PLT transfusion in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to intensive care and receiving at least one platelet transfusion in intensive care unit

Exclusion Criteria:

* Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care and receiving platelet transfusion whatever the reason for it.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
platelet transfusion efficacy | between 18 hours and 28 days after transfusion
  corrected count platelet increment

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU d'Angers, Angers
  - CHRU de Brest, Brest
  - CH des Pays de Morlaix, Morlaix
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes
  - CHU de Tours, Tours
  - Chba Site de Vannes, Vannes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending three years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Derived] Reizine F, Le Marec S, Le Meur A, Consigny M, Berteau F, Bodenes L, Geslain M, McQuilten Z, Le Niger C, Huntzinger J, Seguin P, Thibert JB, Simon D, Reignier J, Egreteau PY, Tadie JM, Huet O, Asfar P, Ehrmann S, Aubron C. Prophylactic platelet transfusion response in critically ill patients: a prospective multicentre observational study. Crit Care. 2023 Sep 27;27(1):373. doi: 10.1186/s13054-023-04650-z. PMID 37759268